CLINICAL TRIAL: NCT03237325
Title: A Pivotal, Double-Blind, Randomized, Placebo-Controlled, Multinational Study of SGX942 (Dusquetide) for the Treatment of Oral Mucositis in Patients Being Treated With Concomitant Chemoradiation for the Treatment of Squamous Cell Carcinoma of the Head and Neck
Brief Title: DOM-INNATE: Study of SGX942 for the Treatment of Oral Mucositis in Patients With Concomitant Chemoradiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDR-OM-02
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Results first posted 2022-08-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity and Oropharynx; Oral Mucositis
Keywords: OM; Head and Neck Cancer; SGX942; Dusquetide; Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Stomatitis; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — dusquetide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGX942 (Experimental): Patients are randomized 1:1 active/placebo.
  Interventions: Drug: SGX942
- Placebo (Placebo Comparator): Patients are randomized 1:1 active/placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGX942 — 1.5 mg/mL SGX942 administered as a 4 minute IV infusion, twice per week starting within 3 days after initiating radiation therapy and continuing through 2 weeks after radiation therapy ends.
  Other Names: Dusquetide
  Arms: SGX942
Drug: Placebo — Placebo is 0.9% sodium chloride (normal saline). The treatment preparation, frequency and duration of therapy are identical to that of the active drug.
  Arms: Placebo

SUMMARY:
To assess the efficacy of SGX942 compared to placebo in decreasing the duration of severe oral mucositis in patients receiving chemoradiation treatment for the treatment of head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven squamous cell carcinoma of the oral cavity or oropharynx without distant organ metastases
* Scheduled to receive cisplatin chemotherapy of 80-100 mg/m²
* Scheduled to receive a continuous course of fractionated, conventional external beam with a cumulative radiation dose between 55 and 72 Gy at each site

Exclusion Criteria:

* Current mucositis
* Current, clinically significant, active infection that in the opinion of the Investigator would make them an unfit participant in the trial
* Planned to receive Erbitux™ (Cetuximab) or similar targeted therapy between Baseline and 6 weeks post-RT
* Prior radiation to the head and neck
* Chemotherapy treatment within the previous 12 months
* Tumors of the lips, sinuses, salivary glands, nasopharynx, hypopharynx, or larynx
* Evidence of significant renal, hepatic, hematologic, or immunologic disease determined by any one of the following: Estimated creatinine clearance <30 mL/min; ALT or AST level greater than 10-fold the upper limit of normal or total bilirubin greater than 3-fold the upper limit of normal; Manifestations of end-stage liver disease, such as ascites or hepatic encephalopathy; Thrombocytopenia; or CD4+ T cell count below 200 cells per μL
* Evidence of immediate life-threatening disease or a life expectancy of less than 3 months
* Women who are pregnant or breast-feeding
* Participation in any study involving administration of an investigational agent within 30 days of randomization into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (53):
- United States (32):
  - Arizona Clinical Research Center, Tucson, Arizona
  - Loma Linda University Health, Loma Linda, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Lakes Research, Miami Lakes, Florida
  - University Cancer & Blood, Athens, Georgia
  - Augusta University, Augusta, Georgia
  - Memorial Health, Savannah, Georgia
  - University of Illinois Cancer Center, Chicago, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ashland Bellefonte Cancer Center, Ashland, Kentucky
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology, Saint Louis Park, Minnesota
  - University of Missouri-Ellis Fischel Cancer Center, Columbia, Missouri
  - Great Falls Clinic, Great Falls, Montana
  - CHI Health St. Francis, Grand Island, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hackensack Meridian Health, Neptune City, New Jersey
  - University of Rochester, Rochester, New York
  - Summa Health Cancer Research, Akron, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Mercy Clinic Oncology and Hematology, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists, Tulsa, Oklahoma
  - Charleston Cancer Center, Charleston, South Carolina
  - Spartanburg Regional-Gibbs Cancer Center, Spartanburg, South Carolina
  - University of Virginia, Charlottesville, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Centre Hospitalier Jolimont, La Louvière
  - Centre Hospitalier Universitaire de Mons, Mons
- France (6):
  - CFRO Clinique Pasteur, Brest
  - Institut Andrée Dutreix, Dunkirk
  - Clinique Victor Hugo, Le Mans
  - Hôpital de la Croix Rousse, Lyon
  - CROM-Osny, Osny
  - Centre Hospitalier Privé St Grégoire, Saint-Grégoire
- Spain (8):
  - Institut Català d'Oncologia Badalona, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia Girona, Girona
  - Hospital Universitario Severo Ochoa, Leganés
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
- United Kingdom (4):
  - Aberdeen Royal Infirmary, Aberdeen
  - Edinburgh Cancer Centre, Edinburgh
  - Guy's Hospital, London
  - Weston Park Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] North JR, Takenaka S, Rozek A, Kielczewska A, Opal S, Morici LA, Finlay BB, Schaber CJ, Straube R, Donini O. A novel approach for emerging and antibiotic resistant infections: Innate defense regulators as an agnostic therapy. J Biotechnol. 2016 May 20;226:24-34. doi: 10.1016/j.jbiotec.2016.03.032. Epub 2016 Mar 23. PMID 27015977
- [Background] Kudrimoti M, Curtis A, Azawi S, Worden F, Katz S, Adkins D, Bonomi M, Elder J, Sonis ST, Straube R, Donini O. Dusquetide: A novel innate defense regulator demonstrating a significant and consistent reduction in the duration of oral mucositis in preclinical data and a randomized, placebo-controlled phase 2a clinical study. J Biotechnol. 2016 Dec 10;239:115-125. doi: 10.1016/j.jbiotec.2016.10.010. Epub 2016 Oct 13. PMID 27746305
- [Background] Kudrimoti M, Curtis A, Azawi S, Worden F, Katz S, Adkins D, Bonomi M, Scott Z, Elder J, Sonis ST, Straube R, Donini O. Dusquetide: Reduction in oral mucositis associated with enduring ancillary benefits in tumor resolution and decreased mortality in head and neck cancer patients. Biotechnol Rep (Amst). 2017 May 17;15:24-26. doi: 10.1016/j.btre.2017.05.002. eCollection 2017 Sep. PMID 28649557

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SGX942 | Placebo
Started | 127 | 139
Completed | 112 | 114
Not Completed | 15 | 25
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 2 | 4
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Noncompliance with Study Procedures | 1 | 1
Not completed — Termination by Sponsor | 0 | 1
Not completed — Reason other than described | 0 | 2

BASELINE CHARACTERISTICS:
Population: The baseline analysis population was defined as all participants that were treated with at least one dose of treatment (SGX942 or Placebo)
Groups:
- Total: Total of all reporting groups
Arm/Group | SGX942 | Placebo | Total
Number analyzed (Participants) | 127 | 139 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (7.48) | 58.8 (8.74) | 58.1 (8.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 28 | 50
  Male | 105 | 111 | 216
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 15 | 24
  Not Hispanic or Latino | 105 | 113 | 218
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 118 | 128 | 246
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
HPV Status [Count of Participants; unit: Participants]
  Positive | 93 | 92 | 185
  Negative | 34 | 47 | 81

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Oral Mucositis (SOM)
Description: To assess the efficacy of SGX942 compared to placebo in decreasing the duration of severe oral mucositis (SOM; defined as World Health Organization [WHO] Grade ≥3). Duration of SOM is defined as the number of days from the onset of SOM until resolution of SOM. OM is evaluated using the published WHO OM grading scale that uses a scale of 0 to 4, with SOM defined as a score ≥3.
Time Frame: approx. 13 weeks
Population: The analysis population was defined as all participants receiving a minimum of 55 Gray of cumulative radiation.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SGX942 | Placebo
Number analyzed (Participants) | 118 | 130
days | 12.5 [4.0 to 22.0] | 20.0 [12.0 to 29.0]
Statistical Analysis 1: Comparison: SGX942 vs Placebo; Test type: Superiority; p = 0.1798, Log Rank

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected between randomization through 6 weeks after radiation therapy treatment ended. Participants received up to 7 weeks of radiation, for a maximum AE collection time of 13 weeks.
Arm/Group | SGX942 | Placebo
All-Cause Mortality (participants affected / at risk) | 7/127 | 9/139
Serious Adverse Events (participants affected / at risk) | 74/127 | 64/139
Other Adverse Events (participants affected / at risk) | 123/127 | 135/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SGX942 (N=127) | Placebo (N=139)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 3
Dysphagia (Gastrointestinal disorders) | 5 | 5
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 4
Oral pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Death (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 3
Bronchiolitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 3 | 1
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 4
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 12 | 8
Renal failure (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Embolism (Vascular disorders) | 4 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SGX942 (N=127) | Placebo (N=139)
Anaemia (Blood and lymphatic system disorders) | 20 | 31
Neutropenia (Blood and lymphatic system disorders) | 21 | 16
Deafness (Ear and labyrinth disorders) | 8 | 7
Hypoacusis (Ear and labyrinth disorders) | 7 | 8
Tinnitus (Ear and labyrinth disorders) | 29 | 37
Constipation (Gastrointestinal disorders) | 71 | 66
Diarrhoea (Gastrointestinal disorders) | 32 | 34
Dry mouth (Gastrointestinal disorders) | 61 | 68
Dyspepsia (Gastrointestinal disorders) | 20 | 23
Dysphagia (Gastrointestinal disorders) | 55 | 60
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 10
Nausea (Gastrointestinal disorders) | 88 | 97
Odynophagia (Gastrointestinal disorders) | 17 | 12
Oesophagitis (Gastrointestinal disorders) | 7 | 7
Oral pain (Gastrointestinal disorders) | 20 | 21
Salivary duct inflammation (Gastrointestinal disorders) | 7 | 4
Stomatitis (Gastrointestinal disorders) | 9 | 21
Vomiting (Gastrointestinal disorders) | 43 | 57
Asthenia (General disorders) | 17 | 11
Chills (General disorders) | 7 | 2
Fatigue (General disorders) | 57 | 64
Medical device site pain (General disorders) | 8 | 6
Pyrexia (General disorders) | 17 | 13
Candida infection (Infections and infestations) | 20 | 20
Oral candidiasis (General disorders) | 34 | 40
Radiation skin injury (Injury, poisoning and procedural complications) | 46 | 55
Alanine aminotransferase increased (Investigations) | 4 | 9
Blood creatinine increased (Investigations) | 14 | 21
Blood urea increased (Investigations) | 8 | 4
Lymphocyte count decreased (Investigations) | 6 | 9
Neutrophil count decreased (Investigations) | 12 | 17
Weight decreased (Investigations) | 32 | 34
White blood cell count decreased (Investigations) | 8 | 14
Decreased appetite (Metabolism and nutrition disorders) | 38 | 43
Dehydration (Metabolism and nutrition disorders) | 26 | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 23 | 23
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Dizziness (Nervous system disorders) | 27 | 17
Dysgeusia (Nervous system disorders) | 58 | 61
Headache (Nervous system disorders) | 31 | 23
Somnolence (Nervous system disorders) | 9 | 8
Anxiety (Psychiatric disorders) | 12 | 15
Depression (Psychiatric disorders) | 4 | 8
Insomnia (Psychiatric disorders) | 14 | 21
Acute kidney injury (Renal and urinary disorders) | 13 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 16
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 18 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 40 | 44
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 11
Erythema (Skin and subcutaneous tissue disorders) | 8 | 13
Rash (Skin and subcutaneous tissue disorders) | 7 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 9 | 5
Hypertension (Vascular disorders) | 4 | 16
Hypotension (Vascular disorders) | 10 | 10
Lymphoedema (Vascular disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03237325/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT03237325/SAP_003.pdf